CLINICAL TRIAL: NCT01120938
Title: Do Pacifiers Protect From Sudden Infant Death Syndrome (SIDS) Through an Increase in Upper Airway Patency?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Israel Amirav MD, Ziv Medical center
Other Study IDs: 07-09
Record Dates: First submitted 2010-05-08; First posted 2010-05-11 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Sudden Infant Death
Keywords: AIrways, Patency, Infant death
MeSH Terms: conditions — Sudden Infant Death; Infant Death

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sudden infant death syndrome (SIDS) is the leading cause of death among infants between 1 month and 1 year of age in the developed world. SIDS continues to be a phenomenon of unknown cause. The best approach to for prevention in high risk infants is unclear. Several substantial lines of evidence indicate that pacifiers have a protective effect on the incidence of SIDS. These studies were significantly powered and the results were consistent world-wide. The explanation for the protective effects of pacifiers on SIDS prevalence is unclear. A recent case report from New Zealand showed by means of nasopharyngeal films of a baby with and without a pacifier the possibility that sucking on a pacifier is associated with a forward movement of the tongue with enlargement of the upper airways' cross sectional area. Indeed, this hypothesis was originally postulated 30 years ago by Cozzi et al.

Working hypothesis and aims: Our hypothesis is that since the upper respiratory tract is that portion of the airway that imposes the greatest resistance to ventilation, sucking on a pacifier results in upper airway dilatation, thus greatly reducing upper airway obstruction and improving ventilation at a stage when infants are virtually obligate nasal breathers. It should be stressed that airway resistance is proportional to the 3rd power of the radius of the airway, thus even a relatively small increase in airway diameter may have a profound effect on airway resistance and respiratory mechanical work of breathing! In young infants and those with underdeveloped respiratory center drive, this decrease in the work of breathing could certainly be sufficient to minimize the risk of SIDS as described above.Thus, the aim of this study is to demonstrate the effect of sucking on a pacifier on upper airway patency.

DETAILED DESCRIPTION:
Ten to 12 infants' parents who have been referred for clinical examination of MR (or CT with and without contrast) of the brain and neck and who require sedation to perform this examination will be asked to participate in the study. These infants represent a potentially ideal population in which to study the upper airway. They are already undergoing MR/CT, their upper airways images are recorded, are asleep, and do not typically have airway abnormalities. In these children, 2 images of the upper airways -one obtained while with and one obtained while without a pacifier -will be analyzed and compared. In no case will additional sedation be given to obtain the MR/CT images of the airway. If the patient begins to wake up during the investigational sequence, the sequence will be aborted.

To test our hypothesis using the functional method, we will compare LRT aerosol penetration with and without a pacifier.

Infants who are regular pacifier users and are receiving therapeutic aerosols regularly (e.g., ventolin, budicort) will be studied. Labeling the aerosol particles with a gamma emitting isotope marker and quantifying its deposition scintigraphically by means of a gamma camera is a simple, safe and commonly used method to assess aerosol deposition throughout the URT and LRT.

ELIGIBILITY:
Inclusion Criteria:

-Infants who have been referred for clinical examination of MR (or CT with and without contrast) of the brain and neck -

* Regular (at least 2 hours a day) of a pacifier

Exclusion Criteria:

-Infants who have histories and/or signs, or symptoms of airway abnormalities -

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Upper airway caliber and patency | 10-20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Israel Amirav, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- Ziv Medical center, Safed, Israel

REFERENCES:
- [Derived] Amirav I, Newhouse MT, Luder A, Halamish A, Omar H, Gorenberg M. Feasibility of aerosol drug delivery to sleeping infants: a prospective observational study. BMJ Open. 2014 Mar 26;4(3):e004124. doi: 10.1136/bmjopen-2013-004124. PMID 24670428